CLINICAL TRIAL: NCT05489861
Title: The Effect of Affirmation and Massage on Babies on Sleep Quality and Maternal-Paternal Attachment: Randomized Controlled Experimental Study
Brief Title: The Effect of Affirmation and Massage on Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Şener Özovalı, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUC-NilaySener
Record Dates: First submitted 2022-07-18; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Attachment; Mother-Infant Interaction; Sleep Quality
Keywords: Baby massage; mother-baby attachment; father-baby attachment; affirmation; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group A The Group to which the Mother Applies Affirmation and Massage (Experimental): 15 minutes of affirmation and massage practices, 3 days a week for 5 weeks, will be taught.
  Affirmation and massage practices will be shown once in the practice hall of the center as an example for the mother to apply to their baby.
  Afterward, affirmation and massage applications will be applied by the mother and father at the baby's home.
  Parents will be informed about the importance of having the same characteristics of the practice room for each application.
  In addition, the massage video material will be given to the mother with an affirmation note as a reminder.
  Interventions: Behavioral: M-AM
- Experimental group B The Group to which the Father Applies Affirmation and Massage (Experimental): 15 minutes of affirmation and massage practices, 3 days a week for 5 weeks, will be taught.
  Affirmation and massage practices will be shown once in the practice hall of the center as an example for the father to apply to their baby.
  Afterward, affirmation and massage applications will be applied by the mother and father at the baby's home.
  Parents will be informed about the importance of having the same characteristics of the practice room for each application.
  In addition, the massage video material will be given to the father with an affirmation note as a reminder.
  Interventions: Behavioral: F-AM
- Control Group (C) (No Intervention): Parents will be asked to continue the implementation of routine sleeping techniques without being taught any practices.

INTERVENTIONS:
Behavioral: M-AM — To examine the effects of affirmation and infant massage taught to their parents on their infants' sleep quality and parent-infant attachment.
  Arms: Experimental group A The Group to which the Mother Applies Affirmation and Massage
Behavioral: F-AM — To examine the effects of affirmation and infant massage taught to their parents on their infants' sleep quality and parent-infant attachment.
  Arms: Experimental group B The Group to which the Father Applies Affirmation and Massage

SUMMARY:
The research was designed as a randomized controlled trial model to examine the effects of affirmation and infant massage taught to the parents of 0-6 month-old infants registered in a Family Health Center and a Private Medical Center in Istanbul, on the sleep quality of their infants and mother-father-infant attachment. The research will be carried out between August and October 2022 by including the parents of the babies in the scope of the study. The Mother-Father and Infant Information Form and the Extended Infant Short Sleep Questionnaire, the Maternal Attachment Scale, and the Father-Infant Attachment Scale will be used to collect the data.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled experimental study with the aim of examining the effect of affirmation and massage applied by mothers and fathers to their infants on their infants' sleep quality and maternal-paternal attachment. Infants aged 0-6 months will be included in the study. In the study, 15 babies (d=0.80, G=0.80, p=0.05) will be randomly selected for each group, Experimental Group 1: The Group To which the Mother Applies Affirmation and Massage (A), Experimental Group 2: The Group To which the Father Applies Affirmation and Massage (B) and Control Group (C) will be determined as three groups. Some criteria will be considered in infants selected and not selected into groups.

Experimental Group 1: Mothers in Group (A) Affirmation and Massage, Experimental Group 2: Fathers in Group (B) Affirmation and Massage, 3 days a week for 15 minutes, will be taught to apply affirmation and massage. Affirmation and massage applications will be shown once in the practice hall of the center as an example for the mother and father to be applied to their baby. Afterwards, affirmation and massage applications will be applied by the mother and father at the baby's home. After 5 weeks, the experimental and control groups will be invited to the center and the results will be compared by measuring with the data collection tools again.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants
* Non-pregnant mothers
* Mothers and fathers who agree to participate in the study
* Who do not have communication problems
* Who does not have a chronic and mental disease

Exclusion Criteria:

* Babies with any disease
* Diagnosed with sleep a disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Examining the infant's sleep quality of infant massage and affirmation | 1. week
  The extended Infant Short Sleep Questionnaire will be used. At the beginning and end of the research. The survey has no minimum and maximum points. The questionnaire has 13 items based on parents' reports of the baby's sleep patterns.
Examining the infant's sleep quality of infant massage and affirmation | 5. week
  The extended Infant Short Sleep Questionnaire will be used. At the beginning and end of the research. It will apply to both mothers and fathers. This scale does not have a score. The questionnaire has 13 items based on parents' reports of the baby's sleep patterns.
Effect on maternal attachment | 1. weeks
  The Maternal Attachment Inventory will be used. At the beginning and end of the research. Cronbach's alpha values are 0.77 in the first month and 0.82 in the 4th month for mothers. It will only apply to mothers. It is a 26-item scale. this scale's high point is 104 and the low point is 98. A high score on the scale indicates high maternal attachment.
Effect on maternal attachment | 5. weeks
  The Maternal Attachment Inventory will be used. At the beginning and end of the research. Cronbach's alpha values are 0.77 in the first month and 0.82 in the 4th month for mothers. It will only apply to mothers. It is a 26-item scale. this scale's high point is 104 and the low point is 98. A high score on the scale indicates high maternal attachment
Effect on paternal attachment | 1. week
  The paternal-infant attachment scale will be used. At the beginning and end of the research. Higher scores indicate higher attachment. It will only apply to fathers. It is a 19-item scale. Each item of the scale is scored between one and five points. this scale's high point is 90 and the low point is 18. Higher scores indicate higher attachment.
Effect on paternal attachment | 5. weeks
  The paternal-infant attachment scale will be used. At the beginning and end of the research. It will only apply to fathers. It is a 19-item scale. this scale's high point is 90 and the low point is 18. Each item of the scale is scored between one and five points. Higher scores indicate higher attachment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nilay Şener Özovalı, Kadıköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No